CLINICAL TRIAL: NCT00005512
Title: Genetic Epidemiology--Development of Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5030; R01HL060688 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Hypertension; Obesity; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Obesity; Heart Diseases

SUMMARY:
To determine how genetic and environmental factors influence the co-occurrence of obesity and hypertension during development and to identify cardiovascular risk factors in adolescence that will predict cardiovascular disease in adults.

DETAILED DESCRIPTION:
BACKGROUND:

Obesity and hypertension are two of the major risk factors for cardiovascular disease (CVD) and those with obesity have a greater risk of hypertension. In children and adolescents, high body mass index correlates with elevated blood pressure. Genetic factors make a significant contribution to the variation of obesity and hypertension.

DESIGN NARRATIVE:

Anthropometric, cardiovascular, physiologic and physical fitness data were used to investigate a series of critical issues about the etiology, heterogeneity, comorbidity and developmental trajectories of CVD risk factors, including obesity, hypertension and cardiovascular health. Using the two datasets, the main questions of the study were addressed. How do genes and environment act and interact to create covariation between obesity and hypertension, and were the genetic and environmental factors the same at all ages (from childhood to late adolescence and adulthood) in both sexes? Areas of research included the following: causes of individual differences in anthropometric and cardiovascular characteristics, their covariation and developmental change or continuity in adolescence, parent-offspring transmission, prediction of cardiovascular risk, and sex, race and population differences in genetic and environmental contributions on cardiovascular risk factors.

ELIGIBILITY:
No eligibility criteria

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1998-08; Study Completion 2002-07

CONTACTS AND LOCATIONS:
Overall Officials: Hermine Maes — Virginia Commonwealth University

REFERENCES:
- [Background] Beunen G, Thomis M, Maes HH, Loos R, Malina RM, Claessens AL, Vlietinck R. Genetic variance of adolescent growth in stature. Ann Hum Biol. 2000 Mar-Apr;27(2):173-86. doi: 10.1080/030144600282280. PMID 10768422
- [Background] Sicherer SH, Furlong TJ, Maes HH, Desnick RJ, Sampson HA, Gelb BD. Genetics of peanut allergy: a twin study. J Allergy Clin Immunol. 2000 Jul;106(1 Pt 1):53-6. doi: 10.1067/mai.2000.108105. PMID 10887305